CLINICAL TRIAL: NCT06244732
Title: Post-Operative Pain Control After Aortic EndoaneurYsmEctomy
Brief Title: Pain Control After Aortic EndoaneurYsmEctomy (POPEYE)
Acronym: POPEYE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Daniela Mazzaccaro, Co-Investigator, Vascular Surgeon, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POPEYE_CET 131-2023
Record Dates: First submitted 2024-01-27; First posted 2024-02-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Pain, Postoperative; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSB (Experimental): In patients in the RSB Group, repeated blocks of the abdominal wall will be performed using special catheters positioned bilaterally in the rectus muscle fascia using ultrasound guidance (Ropivacaine 0.375% 20 ml per side, administered every 12 hours: at T0, T12 and T24)
  Interventions: Procedure: Postoperative pain control
- EA (Active Comparator): Patients of EA Group will receive analgesia via epidural catheter (Ropivacaine 0.15% with double initial bolus and subsequent continuous infusion 5 ml/h via elastomeric pump)
  Interventions: Procedure: Postoperative pain control

INTERVENTIONS:
Procedure: Postoperative pain control — Postoperative analgesia after OR-AAA

SUMMARY:
Open abdominal aortic aneurysm repair (OR-AAA) is an operation associated with high morbidity, and has 30-day mortality rates of between 4 and 14%. Post-operative pain management represents a primary anesthetic focus.

A better analgesia, in addition to being desirable for the patient, can potentially reduce complications associated with postoperative pain and ensure faster functional recovery.

The modern concept of multimodal analgesia involves the association of multiple drugs and/or analgesic techniques to maximize the quality of analgesia and reduce the side effects of the individual methods. In this context, the addition of epidural analgesia (EA) to the intravenous administration of "traditional" analgesic drugs has assumed the role of gold standard in many surgeries, including OR-AAA.

Over time, EA has proven to be a better analgesic technique than the use of intravenous opioids alone, however there is much uncertainty regarding its ability to reduce complications, morbidity and mortality of patients.

For some time, efforts to research effective, less invasive and safe anesthetic alternatives, have been directed towards the development of multimodal analgesia protocols with the aim of reducing complications and ensuring faster recovery. New approaches to post-operative pain management are emerging, including rectus sheat block (RSB).

Currently there is no evidence regarding the effectiveness of RSB in pain control after OR-AAA.

In this context, the study aims to compare two different post-operative pain management protocols, with the aim of verifying whether the use of RSB can guarantee a non-inferior level of analgesia with reduction of complications compared to AE.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled, single-centre, non-profit, spontaneous study, which involves the evaluation of the control of post-operative pain in a population of adult patients admitted to the General Intensive Care Unit after elective open endoaneurysmectomy of the abdominal aorta.

The study will be conducted by analyzing two groups of patients, randomized to receive ether postoperative analgesia via epidural catheter (EA Group) or repeated blocks of the rectus fascia (RSB Group).

Pre- and intra-operative management In EA Group the epidural catheter will be positioned, according to the normal practices of the Operating Unit, before the operation. The insertion of the catheter will be carried out at the T10-T12 level for a maximum of 5-7 cm in the epidural space.

For both groups under study, the operation will be conducted under balanced general anesthesia, using a volatile anesthetic (Desflurane or Sevoflurane) associated with Remifentanil, with titratable doses in order to guarantee an adequate depth of anesthesia, understood as bispectral index (BIS ) between 40 and 60. Myoresolution will be maintained with the use of neuromuscular monitoring (TOF, Train Of Four).

After intubation, the bladder catheter, nasogastric tube, central venous catheter (with ultrasound-guided technique) will be positioned and the following will be prepared:

* Cell saver for blood recovery
* Body temperature monitoring via throat probe
* Minimally invasive arterial hemodynamic monitoring with FloTrac system and continuous detection of the following parameters:

  * Mean arterial pressure (MAP)
  * Cardiac Index (CI)
  * Stroke Volume Variation (SVV) These parameters, as usual, will guide the anesthetic conduct for the optimization of blood volume and intraoperative hemodynamic performance.
* Prophylaxis of nausea and vomiting will be carried out by administering Dexamethasone 4 mg to all patients at induction and Ondansetron 4 mg before extubation
* Upon closure of the abdominal muscle fascia, intravenous analgesia will be administered with Paracetamol 1 g, Ibuprofen 600 mg and MgSO4 2 g At the end of the surgical procedure, each patient, as usual and regardless of the study protocol, will be transferred to the General Intensive Care Unit, where monitoring and the subsequent recovery phase will continue.

Post-operative management All patients will be transferred to the General Intensive Care Unit with continued sedation and mechanical ventilation, in order to standardize the close monitoring of vital functions, the recovery phase and the management of the analgesia protocol.

Each patient will be eligible for awakening and extubation - and therefore for the start of the analgesia protocol - once all the following criteria have been met:

* Body temperature ≥ 35.5° C
* MAP ≥ 65 mmHg (with max basic norepinephrine dosage 0.1 mcg/kg/min)
* TOF-Ratio ≥ 0.9 If the conditions for awakening are not respected, the clinical conditions will be optimized in order to restore the stability necessary for extubation. Patients who have not reached the aforementioned criteria within 12 hours of admission to the ICU will exit the study protocol (see "drop-out criteria").

From the moment of awakening (T0), observation and data collection will continue in the Intensive Care Unit for a total of 36 hours.

Analgesia protocol

The administration of analgesia according to the usual protocols will begin before awakening in those patients who have met the criteria for extubation:

* Group EA will receive analgesia via epidural catheter (Ropivacaine 0.15% with double initial bolus and subsequent continuous infusion 5 ml/h via elastomeric pump)
* in the RSB Group, repeated blocks of the abdominal wall will be performed using special catheters positioned bilaterally in the rectus muscle fascia using ultrasound guidance (Ropivacaine 0.375% 20 ml per side, administered every 12 hours: at T0, T12 and T24) In addition, both groups will be administered intravenous analgesia at predetermined times: 1 g of paracetamol QID (quater in day, except for patients <50 kg and/or with risk factors for hepatotoxicity in which it will be administered in a total dose of 3 g/day), 600 mg of ibuprofen BID (bis in day) and 2 g of MgSO4 TID (tris in day).

Pain symptoms will be assessed according to the NRS scale. This system involves the direct evaluation by the patient of the degree of pain perceived on a scale ranging from 0 (no pain) to 10 (worst possible pain). In our study we will consider values greater than or equal to 4 to be unacceptable. In this case, rescue therapy with opioids is envisaged in addition to the intravenous therapy normally administered. The opioid of choice for our protocol is intravenous morphine, administered in boluses at a dosage of 2 mg, repeatable every 15 minutes (= max 8 mg in one hour) until pain symptoms improve with NRS<4 or appearance of side effects, considering a maximum daily dose of 50 mg.

Data collection

The following variables will be collected from the medical records, which will then be pseudonymised and inserted into a database to be adequately analysed:

1. Pre-operative:

   1. Anthropometric parameters (age, sex, BMI)
   2. ASA class
   3. Revised Cardiac Risk Index
   4. METS
   5. Major comorbidities:

   i) Diabetes mellitus (DM) ii) Ischemic heart disease (IC) iii) Heart failure (HFS) iv) Chronic obstructive pulmonary disease (COPD) v) Chronic kidney disease (CKD) vi) Other significant pathologies
2. Intra-operative:

   a) Type of surgical procedure i) aortobisiliac repair (AO-BIS) ii) aorto-bifemoral repair (AO-BIF) iii) aorto-aortic (AO-AO) repair b) Surgical time c) Time and type of aortic clamping d) Hemodynamic parameters and events i) Maximum dosage of Norepinephrine (mcg/kg/min) ii) MAP ≤ 65 mmHg iii) FloTrac: CI ≤ 2 L/min and/or SVV > 13% iv) Water balance v) Total transfusions in ml (exogenous + blood recovery) vi) Intraoperative AAII thrombotic complications
3. Post-operative:

   a) Pain (NRS scale) both at rest ("static") and upon coughing ("dynamic") i) upon awakening (T0) ii) 2, 4, 8, 12, 18, 24, 30, 36 hours after waking up b) Total dose of rescue opioid c) Occurrence of complications related to the operation and/or the patient's comorbidities i) Re-intervention ii) Thrombosis AAII iii) Hemorrhage iv) major cardiac complications (ACS, ACC, arrhythmias) v) infectious complications (wound infection, sepsis, septic shock) vi) pulmonary complications (pneumonia, respiratory failure, pulmonary edema) vii) acute renal failure d) Occurrence of complications related to the therapy administered i) Nausea/vomiting from opioid consumption ii) Failure of the analgesic technique (uncontrolled pain) iii) Hypotension treatable with max norepinephrine base 0.1 mcg/kg/min iv) Hypotension not treatable without higher doses of basic norepinephrine v) Paresthesia of lower limbs vi) Motor deficit of lower limbs vii) Other complications of AE: direct neurological damage, dural puncture headache, subarachnoid injection/spinal anesthesia, urinary retention, low back pain, epidural hematoma, infection, drug allergy, AL absorption viii) Other complications of RSB: infections, fascial hematoma, drug allergy, AL absorption The analysis continues for a total period of 36 hours after waking up in the Intensive Care Unit. The length of in-hospital stay will be also recorded.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age > 18 years)
* patients who have given their consent to participate in the study
* patients undergoing elective "open" surgical treatment of an abdominal aortic aneurysm with a midline xipho-pubic incision.

Exclusion Criteria:

* Pregnant women
* Patients being treated for chronic pain
* Known allergy to drugs included in analgesia protocols
* Contraindications to the use of one of the two methods provided:

  * refusal by the patient
  * infection at the puncture site
  * coagulopathy:

    1. PTT > 40 s and/or INR > 1.4
    2. platelet count < 50,000/µL
    3. taking antiplatelet or anticoagulant drugs that have not been discontinued in good time, according to international guidelines
* Emergent intervention
* Lack of consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain evaluation | day 0 (12 h after extubation)
  Postoperative pain will be evaluated using Numerical Rating Scale (NRS) (from 0 to 10, where 0 indicates no pain and 10 is the worst pain ever had)

SECONDARY OUTCOMES:
Opioids consumption | within 36 hours from extubation
  Quantify and compare the consumption of opioids administered to optimize analgesia ("rescue") in case of uncontrolled pain in the two groups during the observation period
Complications associated to postoperative analgesia | within 36 hours from extubation
  Detect the onset of complications related to the analgesia technique performed in the study groups

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chang DC, Parina RP, Wilson SE. Survival After Endovascular vs Open Aortic Aneurysm Repairs. JAMA Surg. 2015 Dec;150(12):1160-6. doi: 10.1001/jamasurg.2015.2644. PMID 26331571
- [Result] Hicks CW, Wick EC, Canner JK, Black JH 3rd, Arhuidese I, Qazi U, Obeid T, Freischlag JA, Malas MB. Hospital-Level Factors Associated With Mortality After Endovascular and Open Abdominal Aortic Aneurysm Repair. JAMA Surg. 2015 Jul;150(7):632-6. doi: 10.1001/jamasurg.2014.3871. PMID 25970850
- [Result] Deery SE, Schermerhorn ML. Open versus endovascular abdominal aortic aneurysm repair in Medicare beneficiaries. Surgery. 2017 Oct;162(4):721-731. doi: 10.1016/j.surg.2017.01.022. Epub 2017 Mar 23. PMID 28343694
- [Result] Wanhainen A, Verzini F, Van Herzeele I, Allaire E, Bown M, Cohnert T, Dick F, van Herwaarden J, Karkos C, Koelemay M, Kolbel T, Loftus I, Mani K, Melissano G, Powell J, Szeberin Z, Esvs Guidelines Committee, de Borst GJ, Chakfe N, Debus S, Hinchliffe R, Kakkos S, Koncar I, Kolh P, Lindholt JS, de Vega M, Vermassen F, Document Reviewers, Bjorck M, Cheng S, Dalman R, Davidovic L, Donas K, Earnshaw J, Eckstein HH, Golledge J, Haulon S, Mastracci T, Naylor R, Ricco JB, Verhagen H. Editor's Choice - European Society for Vascular Surgery (ESVS) 2019 Clinical Practice Guidelines on the Management of Abdominal Aorto-iliac Artery Aneurysms. Eur J Vasc Endovasc Surg. 2019 Jan;57(1):8-93. doi: 10.1016/j.ejvs.2018.09.020. Epub 2018 Dec 5. No abstract available. PMID 30528142
- [Result] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482
- [Result] Stenger M, Fabrin A, Schmidt H, Greisen J, Erik Mortensen P, Jakobsen CJ. High thoracic epidural analgesia as an adjunct to general anesthesia is associated with better outcome in low-to-moderate risk cardiac surgery patients. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1301-9. doi: 10.1053/j.jvca.2012.12.001. Epub 2013 Jul 29. PMID 23906858
- [Result] Park WY, Thompson JS, Lee KK. Effect of epidural anesthesia and analgesia on perioperative outcome: a randomized, controlled Veterans Affairs cooperative study. Ann Surg. 2001 Oct;234(4):560-9; discussion 569-71. doi: 10.1097/00000658-200110000-00015. PMID 11573049
- [Result] Wijeysundera DN, Beattie WS, Austin PC, Hux JE, Laupacis A. Epidural anaesthesia and survival after intermediate-to-high risk non-cardiac surgery: a population-based cohort study. Lancet. 2008 Aug 16;372(9638):562-9. doi: 10.1016/S0140-6736(08)61121-6. Epub 2008 Aug 8. PMID 18692893
- [Result] Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, Collins KS; MASTER Anaethesia Trial Study Group. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet. 2002 Apr 13;359(9314):1276-82. doi: 10.1016/S0140-6736(02)08266-1. PMID 11965272
- [Result] Ali M, Winter DC, Hanly AM, O'Hagan C, Keaveny J, Broe P. Prospective, randomized, controlled trial of thoracic epidural or patient-controlled opiate analgesia on perioperative quality of life. Br J Anaesth. 2010 Mar;104(3):292-7. doi: 10.1093/bja/aeq006. Epub 2010 Feb 1. PMID 20124282
- [Result] Nishimori M, Low JH, Zheng H, Ballantyne JC. Epidural pain relief versus systemic opioid-based pain relief for abdominal aortic surgery. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD005059. doi: 10.1002/14651858.CD005059.pub3. PMID 22786494
- [Result] Norris EJ, Beattie C, Perler BA, Martinez EA, Meinert CL, Anderson GF, Grass JA, Sakima NT, Gorman R, Achuff SC, Martin BK, Minken SL, Williams GM, Traystman RJ. Double-masked randomized trial comparing alternate combinations of intraoperative anesthesia and postoperative analgesia in abdominal aortic surgery. Anesthesiology. 2001 Nov;95(5):1054-67. doi: 10.1097/00000542-200111000-00006. PMID 11684971
- [Result] Bardia A, Sood A, Mahmood F, Orhurhu V, Mueller A, Montealegre-Gallegos M, Shnider MR, Ultee KH, Schermerhorn ML, Matyal R. Combined Epidural-General Anesthesia vs General Anesthesia Alone for Elective Abdominal Aortic Aneurysm Repair. JAMA Surg. 2016 Dec 1;151(12):1116-1123. doi: 10.1001/jamasurg.2016.2733. PMID 27603002
- [Result] Guay J, Kopp S. Epidural pain relief versus systemic opioid-based pain relief for abdominal aortic surgery. Cochrane Database Syst Rev. 2016 Jan 5;2016(1):CD005059. doi: 10.1002/14651858.CD005059.pub4. PMID 26731032
- [Result] Greco KJ, Brovman EY, Nguyen LL, Urman RD. The Impact of Epidural Analgesia on Perioperative Morbidity or Mortality after Open Abdominal Aortic Aneurysm Repair. Ann Vasc Surg. 2020 Jul;66:44-53. doi: 10.1016/j.avsg.2019.10.054. Epub 2019 Oct 28. PMID 31672606
- [Result] Monaco F, Pieri M, Barucco G, Karpatri V, Redaelli MB, De Luca M, Mattioli C, Bove T, Melissano G, Chiesa R, Landoni G, Zangrillo A. Epidural Analgesia in Open Thoraco-abdominal Aortic Aneurysm Repair. Eur J Vasc Endovasc Surg. 2019 Mar;57(3):360-367. doi: 10.1016/j.ejvs.2018.09.027. Epub 2018 Oct 29. PMID 30385186
- [Result] Salicath JH, Yeoh EC, Bennett MH. Epidural analgesia versus patient-controlled intravenous analgesia for pain following intra-abdominal surgery in adults. Cochrane Database Syst Rev. 2018 Aug 30;8(8):CD010434. doi: 10.1002/14651858.CD010434.pub2. PMID 30161292
- [Result] Dolin SJ, Cashman JN. Tolerability of acute postoperative pain management: nausea, vomiting, sedation, pruritus, and urinary retention. Evidence from published data. Br J Anaesth. 2005 Nov;95(5):584-91. doi: 10.1093/bja/aei227. Epub 2005 Sep 16. PMID 16169893
- [Result] Hakim SM, Narouze S, Shaker NN, Mahran MA. Risk factors for new-onset persistent low-back pain following nonobstetric surgery performed with epidural anesthesia. Reg Anesth Pain Med. 2012 Mar-Apr;37(2):175-82. doi: 10.1097/AAP.0b013e3182411048. PMID 22286517
- [Result] Curatolo M, Scaramozzino P, Venuti FS, Orlando A, Zbinden AM. Factors associated with hypotension and bradycardia after epidural blockade. Anesth Analg. 1996 Nov;83(5):1033-40. doi: 10.1097/00000539-199611000-00023. PMID 8895281
- [Result] Ready LB. Acute pain: lessons learned from 25,000 patients. Reg Anesth Pain Med. 1999 Nov-Dec;24(6):499-505. doi: 10.1016/s1098-7339(99)90038-x. No abstract available. PMID 10588551
- [Result] Tran DQ, Van Zundert TC, Aliste J, Engsusophon P, Finlayson RJ. Primary Failure of Thoracic Epidural Analgesia in Training Centers: The Invisible Elephant? Reg Anesth Pain Med. 2016 May-Jun;41(3):309-13. doi: 10.1097/AAP.0000000000000394. PMID 27035462
- [Result] Dobson SW, Weller RS, Edwards C, Turner JD, Jaffe JD, Reynolds JW, Henshaw DS. A randomized comparison of loss of resistance versus loss of resistance plus electrical stimulation: effect on success of thoracic epidural placement. BMC Anesthesiol. 2022 Feb 9;22(1):43. doi: 10.1186/s12871-022-01584-x. PMID 35139802
- [Result] Kehlet H. Labat lecture 2005: surgical stress and postoperative outcome-from here to where? Reg Anesth Pain Med. 2006 Jan-Feb;31(1):47-52. doi: 10.1016/j.rapm.2005.10.005. No abstract available. PMID 16418025
- [Result] Kuniyoshi H, Yamamoto Y, Kimura S, Hiroe T, Terui T, Kase Y. Comparison of the analgesic effects continuous epidural anesthesia and continuous rectus sheath block in patients undergoing gynecological cancer surgery: a non-inferiority randomized control trial. J Anesth. 2021 Oct;35(5):663-670. doi: 10.1007/s00540-021-02973-1. Epub 2021 Jul 15. PMID 34268624
- [Result] Ferreira-Valente MA, Pais-Ribeiro JL, Jensen MP. Validity of four pain intensity rating scales. Pain. 2011 Oct;152(10):2399-2404. doi: 10.1016/j.pain.2011.07.005. PMID 21856077
- [Result] Kietaibl S, Ferrandis R, Godier A, Llau J, Lobo C, Macfarlane AJ, Schlimp CJ, Vandermeulen E, Volk T, von Heymann C, Wolmarans M, Afshari A. Regional anaesthesia in patients on antithrombotic drugs: Joint ESAIC/ESRA guidelines. Eur J Anaesthesiol. 2022 Feb 1;39(2):100-132. doi: 10.1097/EJA.0000000000001600. PMID 34980845
- [Result] Ball L, Pellerano G, Corsi L, Giudici N, Pellegrino A, Cannata D, Santori G, Palombo D, Pelosi P, Gratarola A. Continuous epidural versus wound infusion plus single morphine bolus as postoperative analgesia in open abdominal aortic aneurysm repair: a randomized non-inferiority trial. Minerva Anestesiol. 2016 Dec;82(12):1296-1305. Epub 2016 Aug 30. PMID 27575452
- [Result] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324